CLINICAL TRIAL: NCT00994851
Title: National Study, Phase III, Parallel, Double Blind, Placebo Comparative and Randomized to Evaluate the Therapeutic Efficacy and Tolerability of the Combination Naturetti® (Cassia Fistula + Senna Alexandrina Miller) in the Chronic Functional Constipation.
Brief Title: Evaluation of Cassia Fistula + Senna Alexandrina Miller in the Chronic Functional Constipation Treatment.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SENCA_L_04746
Record Dates: First submitted 2009-10-13; First posted 2009-10-14 (Estimated); Last update posted 2013-03-29 (Estimated); Status verified 2013-03

CONDITIONS: Constipation
MeSH Terms: conditions — Constipation | interventions — Sennosides

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- SENNA+ CASSIA (Experimental): Daily administration (capsule) of Naturetti (SENNA+ CASSIA) at bedtime, during 30 days
  Interventions: Drug: SENNA+CASSIA
- Placebo (Placebo Comparator): Daily administration (capsule) of placebo at bedtime, during 30 days
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: SENNA+CASSIA — Pharmaceutical form: capsule Route of administration: oral Dose regimen: once a day
  Arms: SENNA+ CASSIA
Drug: placebo — Pharmaceutical form: Capsule Route of administration: oral Dose regimen: once a day
  Arms: Placebo

SUMMARY:
Primary Objective:

To evaluate the clinical efficacy of Naturetti (capsules) , considering the following criteria:

* Evacuation frequency during the treatment and follow-up period
* Consistency of stools during the treatment and follow-up period
* Global evaluation, regarding increase in frequency of evacuation and shape of stools.

Secondary Objective:

* Number of days without evacuation
* Proportion of evacuation with pain
* Proportion of evacuation with strain
* Proportion of evacuation with incomplete sensation
* Proportion of blocked stools
* Proportion of manual maneuvers to facilitate defecation
* Proportion of subjects that adhere to the diet recommended
* Proportion of the patients who have to use rescue medication
* Level of constipation improvement, according to the patient evaluation
* To evaluate clinical tolerability of the study medication by the continuous use
* To evaluate the occurrence of adverse events related to the study drug
* To identify any drug interaction.

ELIGIBILITY:
Inclusion criteria:

* Chronic functional constipation present, diagnosed by Rome III criteria.
* Present in most evacuations intestinal feces classified as Type 1 or 2 by the classification of Bristol.
* Women sexually active and reproductive age, using more than three months effective contraceptive method.
* Concordance, level of education and consciousness enough to cooperate with the completion of all study procedures.
* No contraindication to the use of medication in the study.
* Availability to attend all the visits of the study evaluation.

Exclusion criteria:

* History or presence of neurological disorders and / or metabolism.
* Persons with constipation caused by previous surgery.
* Presence of obstructive lesions in the gastrointestinal tract, including colorectal cancer.
* Irritable bowel syndrome or inflammatory bowel disease.
* Multiple Sclerosis
* Parkinson's disease
* Other abnormalities such as Hirschsprung's disease and Defecation Dissinrgica.
* Heart disease and / or hypertension.
* Continuous use of medication such as analgesics, anti-cholinergic (anti-histamines, antispasmodics, antidepressants, anti-psychotics), supplements with iron or aluminum, Opiates, Anti-hypertensive, CALCIUM CHANNEL BLOCKERS Preganglionic and blockers.
* Use of any other except the laxative rescue medication during the study.
* Subjects who do not confirm the diagnosis of ICFC during Phase I of the study.
* Pregnant or breast-feeding period.
* Laboratory tests outside the normal range, or the result is assessed as clinically significant by the Investigator.
* Body Mass Index (BMI) over 30.
* Participation in another clinical study within 30 days.
* Do not fill the correct Diary
* Any condition that in view of the researcher impossible the Subject to participate in the study.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 96 (Actual)
Dates: Start 2009-09; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Evaluation of the evacuation frequency during the treatment and follow-up period | 30 and 45 days
Evaluation of the stools consistency during the treatment and follow-up period | 30 and 45 days
Global evaluation, regarding increase in frequency of evacuation and shape of stools | 30 and 45 days

SECONDARY OUTCOMES:
Number of days without evacuation | 30 days
Proportion of evacuation with pain | 30 days
Proportion of evacuation with strain | 30 days
Proportion of evacuation with incomplete sensation | 30 days
Proportion of blocked stools | 30 days
Proportion of manual maneuvers to facilitate defecation | 30 days
Proportion of subjects that adhere to the diet recommended | 30 days
Proportion of the patients who have to use rescue medication | 30 days
Level of constipation improvement, according to the patient evaluation | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Jaderson Lima, Study Director, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis Administrative Office, São Paulo, Brazil